CLINICAL TRIAL: NCT06696313
Title: Radiographic Migration Analysis of the Insignia Hip Stem
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Collaborators: Orthopaedic Innovation Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B2024:118
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hip Implant; Hip Replacement in Osteoarthritis Patients; Migration of Implant
Keywords: Insignia; RSA; Total hip replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Insignia (Other): Total hip replacement CT-RSA vs gold standard RSA
  Interventions: Device: Insignia

INTERVENTIONS:
Device: Insignia — * Insignia hip stem
  * Trident hemispherical shell
  * X3 polyethylene liner
  * Metal or ceramic head

SUMMARY:
The purpose of this study is to assess the migration pattern of the Insignia hip stem using radiostereometric analysis (RSA for short) and computed tomography (CT). Only patients with degenerative joint disease requiring primary total hip replacement will be asked to participate. The other purpose is to assess if there are any differences between the gold-standard RSA-measured migration and CT-RSA-measured migration. The clinical outcomes will be measured using joint function and patient satisfaction questionnaires. Approximately thirty patients will be enrolled onto the study.

DETAILED DESCRIPTION:
This is a single-centre, non-randomized, non-controlled trial of patients undergoing primary total hip arthroplasty using the Insignia hip stem. Patients will undergo RSA and CT-RSA imaging and analyses to identify migration of the femoral stem with respect to the adjuvant bone during the first 2 post-operative years.

The primary outcome of this study is to determine if femoral stem stability is achieved between 6-12 month and 12-24 month post-operative intervals.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the hip indicating primary total hip arthroplasty - Aged 21 years or older
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery
* Medical condition with less than 2 years life expectancy
* Overhanging pannus (direct anterior approach)
* Prior surgery of the hip involving implantation of hardware (i.e., hemiarthroplasty, internal fixation, pelvic reconstruction near the acetabulum requiring removal)
* Skin condition on the area of incision
* Multi-level lumbar spine fusion
* Ankylosing spondylolithesis
* Shortening osteotomy through the femur

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Migration | Up to 2 years post-operative
  Quantify migration of the Insignia stem using RSA and CT-RSA

SECONDARY OUTCOMES:
Validation | Up to 2 years post-operative
  Comparison of RSA and CT-RSA using the standard deviation of the mean component migration calculated from examinations.
Early migration | Up to 2 years post-operative
  Quantify early migration of the Trident acetabular cup using RSA
Changes in Oxford-12 Hip Score from baseline(pre-op) to 6-month, 1-year and 2-year | Up to 2 years post-operative
  The Oxford Hip Score (OHS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OHS measures pain and general activities of daily living
Changes in EQ-5D-5L from baseline(pre-op) to 6-month, 1-year and 2-year | Up to 2 years post-operative
  The EuroQol 5D 5L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Changes in Patient Satisfaction (VAS) from baseline(pre-op) to 6-month, 1-year and 2-year | Up to 2 years post-operative
  Evaluate and compare the change from preoperative to 2 years in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (Unsatified) - 100 (Completely Satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Bohm, MD, Principal Investigator — Orthopaedic Innovation Centre
Locations (1):
- Concordia Hip & Knee Institute, Winnipeg, Manitoba, Canada